CLINICAL TRIAL: NCT01438086
Title: A Randomised Trial Evaluating the Safety and Efficacy of a Single Low Dose of Intracoronary Insulin-like Growth Factor-1 Following Percutaneous Coronary Intervention for ST-Elevation Acute Myocardial Infarction (RESUS-AMI)
Brief Title: Evaluation of the Safety and Efficacy of Using Insulin-like Growth Factor-1 in Patients With a Heart Attack
Acronym: RESUS-AMI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Professor Noel Caplice, Professor of Cardiovascular Sciences, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UCC-IGF-001; 2011-000480-27 (EudraCT Number)
Record Dates: First submitted 2011-09-17; First posted 2011-09-21 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Heart Failure; Myocardial Infarction
Keywords: Heart Failure; Myocardial Infarction
MeSH Terms: conditions — Heart Failure; Myocardial Infarction | interventions — mecasermin; Insulin-Like Growth Factor I; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- mecasermin low dose (Active Comparator)
  Interventions: Drug: mecasermin
- mecasermin high dose (Active Comparator)
  Interventions: Drug: mecasermin
- saline placebo (Placebo Comparator)
  Interventions: Drug: 0.9% sodium chloride injection

INTERVENTIONS:
Drug: mecasermin — Intracoronary bolus
  Other Names: rhIGF-1; IGF-1
  Arms: mecasermin low dose
Drug: mecasermin — Intracoronary bolus
  Other Names: rhIGF-1; IGF-1
  Arms: mecasermin high dose
Drug: 0.9% sodium chloride injection — Intracoronary bolus
  Other Names: normal saline
  Arms: saline placebo

SUMMARY:
When a patient has a heart attack, a blockage occurs in a coronary artery that delivers oxygen to the heart muscle. The heart muscle may weaken, causing heart failure. The body naturally makes a protein called insulin-like growth factor-1 (IGF-1) that may protect the heart muscle cells from dying and may prevent heart failure or lessen the damage that occurs. IGF-1 is also available as a drug called mecasermin. In this study, heart attack patients will be given either a dose of mecasermin or a placebo (inactive treatment) after their coronary artery has been opened by a stent. The purpose of the study will be to evaluate the safety of the therapy and to test if the therapy will prevent or lessen heart failure by evaluating a cardiac magnetic resonance imaging (MRI) taken one day and eight weeks after the heart attack.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75
* Presents within 2-12 hours of at least 30 minutes of myocardial ischemic pain
* ECG evidence of myocardial infarction
* Undergoing percutaneous coronary intervention (PCI) for ST-elevation myocardial infarction
* Left ventricular ejection fraction during PCI of 40% or less
* TIMI flow grade 3 in the infarct-related artery following reperfusion and stenting

Exclusion Criteria:

* History of prior myocardial infarction
* Prior history of heart failure, left ventricular dysfunction or cardiomyopathy
* Active or suspected neoplasia
* Known impaired liver function
* Cardiogenic shock
* Estimated glomerular filtration rate < 45 ml/min/1.73m2
* History of hypoglycaemia requiring hospitalisation
* History of primary insulin-like growth factor-1 deficiency or growth hormone disorders
* Contraindication to cardiac magnetic resonance imaging
* Pregnancy or nursing mothers
* Known allergy to study drug or any of its inactive ingredients
* Treatment with another investigational agent within 30 days of enrolment
* Subjects unable or unwilling to comply with follow-up requirements of study
* Subjects unable to provide written informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Serum glucose measurement | 30 minutes after study drug administration
  Safety outcome measure
Percent change in global left ventricular ejection fraction (LVEF) measured by quantitative cardiac magnetic resonance imaging (MRI) | Baseline and 8 weeks
  Efficacy outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Noel Caplice, MB, PhD, Principal Investigator — University College Cork
Locations (2):
- Cork University Hospital, Cork, Ireland
- Leiden University Medical Center, Leiden, Netherlands